CLINICAL TRIAL: NCT01242930
Title: A Phase II Trial to Determine the Effect of Imetelstat (GRN163L) on Patients With Previously Treated Multiple Myeloma
Brief Title: Open Label Study With Imetelstat to Determine Effect of Imetelstat in Patients w/ Previously Treated Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Geron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP14B013
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Myeloma
Keywords: imetelstat; imetelstat sodium; GRN163L; telomerase inhibitor; telomerase inhibition; multiple myeloma; myeloma; myeloma progenitor cells
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — imetelstat; GRN163L peptide; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imetelstat (7.5 mg/kg) (Experimental): Imetelstat (7.5 mg/kg) with or without lenalidomide standard of care
  Interventions: Drug: Imetelstat (7.5 mg/kg); Drug: lenalidomide standard of care
- Imetelstat (9.4 mg/kg) (Experimental): Imetelstat (9.4 mg/kg) with or without lenalidomide standard of care
  Interventions: Drug: lenalidomide standard of care; Drug: Imetelstat (9.4 mg/kg)

INTERVENTIONS:
Drug: Imetelstat (7.5 mg/kg) — Imetelstat 7.5 mg/kg as a 2-hour intravenous infusion (± 10 minutes) on Days 1 and 8 of a 28-day cycle; the Day 8 dose will be omitted in patients with a prior history of bone marrow or stem cell transplant.
  Other Names: GRN163L
  Arms: Imetelstat (7.5 mg/kg)
Drug: lenalidomide standard of care — Patients who are receiving lenalidomide as maintenance therapy upon enrollment as part of their treatment regimen may remain on this therapy during trial participation, provided that they have received this treatment for a minimum of 3 months and demonstrate evidence of stabilization of their response.
  Other Names: Revlimid
Drug: Imetelstat (9.4 mg/kg) — Imetelstat 9.4 mg/kg as a 2-hour intravenous infusion (± 10 minutes) on Days 1 and 8 of a 28-day cycle; the Day 8 dose will be omitted in patients with a prior history of bone marrow or stem cell transplant.
  Other Names: GRN163L
  Arms: Imetelstat (9.4 mg/kg)

SUMMARY:
This is an open label Phase II study to determine the rate of improvement in response of patients with previously treated multiple myeloma to imetelstat alone or in combination with lenalidomide maintenance therapy. This study will include multiple myeloma patients who either have achieved disease stabilization or who have achieved at least a partial response (PR) but failed to achieve a complete response (CR) after cytoreductive therapy for multiple myeloma; ie, have detectable but non-progressing disease and will most likely relapse.

ELIGIBILITY:
Inclusion Criteria:

Willing and able to sign an informed consent Male or female, 18 years or older Confirmed diagnosis of multiple myeloma (secretory disease) by International Myeloma Working Group Diagnostic Criteria

Patients must meet one of the following criteria:

o Previously treated patients with multiple myeloma who achieved at least stable disease but who have failed to achieve a complete response (CR) after a minimum of one cytoreductive therapy for multiple myeloma and have detectable but non-progressing disease. Patients must have received at least one proteasome inhibitor (eg, bortezomib) or one immunomodulatory agent (eg, thalidomide or lenalidomide) or both.

Patients receiving lenalidomide as maintenance therapy may continue to receive this therapy provided that the patient has been on this maintenance therapy for a minimum of 3 months and has evidence of disease stabilization.

Disease stabilization will be defined as an M protein that varies ≤ 25% over the three measurements or remains under 0.5 g/dL whichever is smaller.

ECOG performance status 0-2 Life expectancy ≥ 3 months

Laboratory criteria (within 14 days of first study drug administration):

* ANC ≥ 1000/μL
* Platelet count ≥ 50 x 103/μL (without transfusion support within 2 weeks prior to first study drug administration)
* Hemoglobin ≥ 8.0 g/dL
* Serum creatinine ≤ 3 x the upper limit of normal (ULN)
* AST (SGOT) and ALT (SGPT) ≤ 2.5 x the upper limit of normal (ULN), unless due to disease.

Must have fully recovered from any previous cancer treatments and/or major surgery.

Women of childbearing potential must have a negative serum pregnancy test and agree to use effective birth control (two reliable forms of contraception) during and for at least 12 weeks after the last treatment.

Males must agree to use effective birth control for themselves or their partner during and for 12 weeks after the last treatment with imetelstat. For those patients receiving lenolidomide, males must use latex condom during sexual contact with women of childbearing potential even if they have undergone a successful vasectomy.

Exclusion Criteria:

Women who are pregnant or breast feeding Prior radioimmunotherapy. Known intracranial disease or epidural disease. Patients with lytic lesions of the cranium or spine secondary to myeloma are eligible to enroll.

Clinically significant cardiovascular disease or condition including:

* Congestive heart failure (CHF) requiring therapy
* Need for antiarrhythmic therapy for a ventricular arrhythmia
* Severe conduction disturbance
* Angina pectoris requiring therapy
* Uncontrolled hypertension per the Investigator's discretion
* New York Heart Association Class II, III, or IV cardiovascular disease Active or chronically recurrent bleeding (eg, active peptic ulcer disease) Clinically relevant active infection. Serious co-morbid medical conditions, including cirrhosis and chronic obstructive or chronic restrictive pulmonary disease.

Symptomatic hyperviscosity syndrome. Any other cancer therapy including chemotherapy, monoclonal antibody, signal transduction inhibitor, immunotherapy, glucocorticoid (except topical or as premedication), thalidomide within 3 weeks prior to first study drug administration.

Investigational therapy within 4 weeks prior to first study drug administration.

Major surgery within 4 weeks prior to first study drug administration (central line placement is allowed) Anti-platelet therapy within 2 weeks prior to first study drug administration, other than low dose aspirin prophylaxis therapy.

Full dose anticoagulation. Prophylactic low dose administration for management of IV access devices is allowed.

Known positive serology for human immunodeficiency virus (HIV. Any other severe, acute, or chronic medical or psychiatric condition, laboratory abnormality, or difficulty complying with protocol requirements that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Rate of Improvement in Response | From time of first dose (Cycle 1 day 1) through end of study period (12 mos. after last participant is enrolled)
  To determine the rate of improvement in response in patients with previously treated multiple myeloma following treatment with imetelstat alone or in combination wtih lenalidomide maintenance therapy. Response will be assessed using the International Uniform Response Criteria for Multiple Myeloma (IURCMM).

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | From time of first dose (Cycle 1 day 1) through end of study (12 mos. after last participant is enrolled)
  As assessed from Cycle 1 Day 1 to first evidence of PD as defined by IURCMM, or death, whichever occurs first.
Safety and Tolerability | From time of first dose (Cycle 1 day 1) through end of study (12 mos. after last participant is enrolled)
  The safety and tolerability of imetelstat will be assessed by the incidence, nature, relatedness and severity of adverse events, laboratory abnormalities and vital signs.
  Patients who develop Grade 3 or 4 cytopenias (other than lyphophenia and/or leukopenia alon) will receive addiontal safety monitoring for reversibility.

CONTACTS AND LOCATIONS:
Overall Officials: Ted Shih, PharmD, Study Director — Geron Corporation; Carol Ann Huff, M.D., Principal Investigator — Sidney Kimmel Cancer Center at Johns Hopkins Hospital
Locations (2):
- United States (2):
  - University of Maryland Medical Center - M & S Greenebaum Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Cancer Center Johns Hopkins Hospital, Baltimore, Maryland